CLINICAL TRIAL: NCT01958970
Title: A Randomized, Double-blind, Pilot Study of PINTA 745, an Anti-myostatin Peptibody, in Patients With End Stage Renal Disease Who Require Maintenance Hemodialysis and Have Protein Energy Wasting
Brief Title: Effects of PINTA 745 in End Stage Renal Disease (ESRD) Patients Who Require Hemodialysis and Have Protein Energy Wasting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pinta Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 745-201
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: End Stage Renal Disease; Kidney Disease; Protein Energy Wasting
Keywords: End Stage Renal Disease; ESRD; Maintenance Hemodialysis; Hemodialysis; Dialysis; MHD; Protein Energy Wasting; PEW
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PINTA 745 (Experimental)
  Interventions: Drug: PINTA 745
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PINTA 745 — PINTA 745 will be administered once weekly by IV infusion.
  Cohort dose schedules:
  * 3mg/kg weekly for 12 weeks
  * 3mg/kg for 3 weeks, followed by 1mg/kg for 9 weeks
  * 6mg/kg for 3 weeks, followed by 2mg/kg for 9 weeks
  Arms: PINTA 745
Drug: Placebo — Placebo will be administered once weekly by IV infusion.
  Cohort dose schedules:
  * 3mg/kg weekly for 12 weeks
  * 3mg/kg for 3 weeks, followed by 1mg/kg for 9 weeks
  * 6mg/kg for 3 weeks, followed by 2mg/kg for 9 weeks
  Arms: Placebo

SUMMARY:
This is a pilot study to assess the safety, pharmacokinetics and effectiveness of PINTA 745 or placebo in treating protein energy wasting (PEW) in patients receiving maintenance hemodialysis (MHD).

DETAILED DESCRIPTION:
This is a randomized (participants will be assigned by chance to study treatments), double-blind (participants and study personnel will not know the identity of the study treatments), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study in patients who receive maintenance hemodialysis. Three participants will receive PINTA 745 for every participant that receives placebo. PINTA 745 or placebo will be taken intravenously once per week following dialysis.

The study period will consist of screening, treatment for 12 weeks, and follow up for 8 weeks. Evaluations will be performed to assess the safety, pharmacokinetics (study of what the body does to a drug), pharmacodynamics (study of what a drug does to the body) and effectiveness in treating protein energy wasting (such as increasing muscle size and muscle function) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patient and on outpatient maintenance hemodialysis for ≥ 6 months
* Adequate dialysis with Kt/V ≥ 1.2 on two occasions within 12 weeks of enrollment
* Undergoing dialysis at least 3 times per week, on average
* Serum albumin ≤ 3.8g/dL within 60 days of enrollment
* Able and willing to provide Informed consent

Exclusion Criteria:

* Presence of an indwelling central vascular catheter
* Current medical condition that would interfere with ability to perform physical function tests
* Active infection requiring hospitalization or antibiotics within the past month
* Major surgery within past 3 months, minor surgery within the past 4 months
* Dialysis access revision/angioplasty/replacement within the past 2 weeks
* History of renal transplant, whether or not functional, within 2 years (however, if graft has been removed, patient will be considered eligible) or plans to undergo renal transplantation within 6 months
* History of neoplasia, except non-melanoma skin cancers, with a 30% probability of recurrence within 12 months
* Current treatment with appetite stimulants, anabolic steroids or growth hormone
* Clinically significant heart disease
* Difficulty swallowing food or liquid
* If female, currently breast feeding
* If female, pregnant
* If female or male, unwilling to use a highly effective method of contraception

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Percent Changes in Lean Body Mass (LBM) | MTD will be assessed after the last patient in Cohort 1A and Cohort 2A complete 28 days on treatment. LBM will be assessed for comparing baseline to Week 12
  To evaluate the safety, dose-limiting toxicities (DLTs), maximum tolerated dose (MTD) and pharmacokinetics of PINTA 745 and to evaluate percentage change in LBM relative to baseline at 12 weeks, via dual-energy x-ray absorptiometry(DXA) scans, in the group receiving PINTA 745 at the MTD (or if no MTD is reached, at the recommended phase 2 dose)

SECONDARY OUTCOMES:
Change in Muscle Composition - Lean Body Mass (LBM), Appendicular Lean Mass (ALM) and Mid Upper Arm Muscle Circumference (MUAMC) | Baseline through Week 20
  To evaluate the change in LBM and ALM via CT and dual-energy x-ray absorptiometry (DXA) scans relative to baseline at 12, 16 and 20 weeks. To evaluate change relative to baseline in MUAMC at 5, 9, 16 and 20 weeks.
Change in Physical Function | Baseline through Week 20
  To evaluate change in physical function as measured by the Stair Climbing Power Test (SCPT) and the 6 Minute Walk Test (6MWT) relative to baseline at 5, 9, 12, 16 and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Haqq, MD, PhD, Study Director — Pinta Biotherapeutics
Locations (6):
- United States (6):
  - DaVita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - University of Washington, Seattle, Washington